CLINICAL TRIAL: NCT02009046
Title: Randomized Evaluation of a Multi-Component, Rights-Based Sexuality Education Initiative for High School Students
Acronym: SEI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Public Health Institute, California (Other)
Collaborators: University of Southern California (Other); Planned Parenthood Los Angeles (Unknown); Ford Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 04704-01-01
Record Dates: First submitted 2013-11-18; First posted 2013-12-11 (Estimated); Results first posted 2018-10-19 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Pregnancy; Sexually Transmitted Diseases
Keywords: Adolescent; Sex education; Sexuality education; Sexually transmitted diseases; Pregnancy; Sexual behavior; Sexuality; Relationship rights; Gender norms; Human rights; Intervention studies; Parent intervention; Peer intervention
MeSH Terms: conditions — Sexually Transmitted Diseases; Sexual Behavior; Sexuality

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- SEI Classroom Curriculum (Experimental): Participants receive the SEI classroom curriculum.
  Interventions: Behavioral: SEI Classroom Curriculum
- Control Classroom Curriculum (Active Comparator): Participants receive the control classroom curriculum.
  Interventions: Behavioral: Control Classroom Curriculum
- SEI Curriculum + 3 School Components (Experimental): Participants receive SEI classroom curriculum and three school wide components (peer advocacy and education, parent education, clinical services linkages).
  Interventions: Behavioral: SEI Curriculum + 3 School Components
- Control Curriculum + 1 School Component (Active Comparator): Participants receive control classroom curriculum and one of the three school wide components (clinical services linkages).
  Interventions: Behavioral: Control Curriculum + 1 School Component

INTERVENTIONS:
Behavioral: SEI Classroom Curriculum — Participants receive the 12-session Sexuality Education Initiative (SEI) classroom curriculum. The SEI classroom curriculum covers anatomy, abstinence, contraception and protection, STIs and HIV/AIDS, media messages, gender, relationships, rights and responsibilities, pregnancy, sexuality, peer pressure, negotiation and coercion, and decision making. These sessions are delivered over a two-month period. Each curriculum session is about 45 minutes in length.
  Arms: SEI Classroom Curriculum
Behavioral: Control Classroom Curriculum — Participants receive the 3-session basic control curriculum. The control curriculum includes 3 sessions on sexually transmitted infections, anatomy and birth control delivered over a two- or three-week period. Each curriculum session is about 45 minutes in length.
  Arms: Control Classroom Curriculum
Behavioral: SEI Curriculum + 3 School Components — Participants receive SEI classroom curriculum and all three school wide components. The peer education/advocacy component recruits, trains and supervises students through an after-school leadership program to serve as resources to peers, organize health events, and refer students to school-based clinic services. The parent education component provides sessions for parents of students, covering reproductive health, teen pregnancy, and parent-teen communication, together with a parent education booklet for widespread use. The clinical services linkages includes health services on campus, including pregnancy/STI testing, contraceptive consultation and prescriptions, condom distribution, counseling, and referrals. It includes training for teachers and staff to distribute condoms as needed.
  Arms: SEI Curriculum + 3 School Components
Behavioral: Control Curriculum + 1 School Component — Participants receive control classroom curriculum and one of the three school wide components, the clinical services linkages. This component includes health services on campus for students, including pregnancy and STI testing, contraceptive consultation and prescriptions, condom distribution, counseling, and referrals. It also includes training for teachers and school staff to distribute condoms to students as needed.
  Arms: Control Curriculum + 1 School Component

SUMMARY:
This study examines the effectiveness of the Sexuality Education Initiative (SEI), a comprehensive, multi-component, rights-based sexuality education program developed and implemented by Planned Parenthood Los Angeles for high school students. The primary goal of the SEI is to improve the sexual and reproductive health of youth attending Los Angeles high schools. The SEI consists of four intervention components: (1) a 12-session gender-sensitive, rights-based, comprehensive sexuality education curriculum, (2) a peer education and advocacy component, (3) a parent education component, and (4) clinical services linkages. It is hypothesized that the 12-session classroom curriculum is more effective than a 3-session control sex education curriculum. It is also hypothesized that the full SEI package (all four components) is more effective than the control condition (control curriculum and clinical services only).

DETAILED DESCRIPTION:
This study examines the effectiveness of the Sexuality Education Initiative (SEI), a comprehensive, multi-component, rights-based sexuality education program developed and implemented by Planned Parenthood Los Angeles for high school students. The primary goal of the SEI is to improve the sexual and reproductive health of youth attending Los Angeles high schools. The SEI consists of four intervention components: (1) a 12-session gender-sensitive, rights-based, comprehensive sexuality education curriculum, (2) a peer education and advocacy component, (3) a parent education component, and (4) clinical services linkages.

* The 12-session gender-sensitive, rights-based classroom curriculum covers anatomy, abstinence, contraception and protection, STIs and HIV/AIDS, media messages, gender, relationships, rights and responsibilities, pregnancy, sexuality, peer pressure, negotiation and coercion, and decision making.
* The peer education and advocacy component recruits, trains and supervises students through an after-school leadership program to serve as school-wide resources to their peers, organize health events at school, and refer students to school-based clinic services.
* The parent education component consists of a series of sessions for parents, covering reproductive health, teen pregnancy, and parent-teen communication, together with a parent education booklet for widespread use.
* The in-school clinical services component provides "clinic without walls" health services on campus, including pregnancy and STI testing, contraceptive consultation and prescriptions, condom distribution, counseling, and referrals. It also trains teachers and school staff to distribute condoms to students as needed.

The evaluation design involves two levels of randomization: First, all schools are randomized into one of two conditions: receiving all three SEI school wide components (peer, parent, clinical services) or receiving only one of these three school wide components (clinical services). Schools are randomized within matched pairs of demographically similar schools. Second, within each school, classrooms are randomized into one of two conditions: a basic 3-session sex education curriculum (control) or the 12-session SEI curriculum (intervention). Thus, all participating 9th grade students will receive at least three sexuality education curriculum sessions and access to on-site clinic services.

The primary research questions for the evaluation are:

1. Is the 12-session SEI gender-sensitive, rights-based sexuality education curriculum more effective than a 3-session comparison curriculum in reducing risk of unwanted pregnancy and sexually transmitted infections (STIs) among high school students?
2. Is the full comprehensive program (all four components as a package) more effective than the two-component comparison condition (only the 3-session comparison curriculum and the clinical services linkages) in reducing risk of teen pregnancies and STIs?

The first hypothesis is that the 12-session SEI gender-sensitive, rights-based curriculum is more effective than the 3-session comparison curriculum in improving sexual health outcomes (as defined in section 7) among program participants one year after participation in the program. The second hypothesis is that the full SEI program (all four components as a package) is more effective than the comparison condition (only the 3-session comparison curriculum and the clinical services linkages) in improving sexual health outcomes one year after participation.

In addition to addressing these questions using the designated primary and secondary outcomes, this study will examine changes in the following short-term outcomes that measure critical concepts being addressed by the curriculum and serve as the hypothesized mediators in the SEI theory of change:

* Attitudes about rights in sexual relationships
* Communication about relationships, rights and sexuality with partners
* Communication about relationships, rights and sexuality with parents/ guardians
* Access to accurate information about sexuality and sexual health
* Knowledge about sex, sexuality and sexual risk protection
* Self-efficacy to assert sexual limits and manage risky situations
* Intentions to protect self from sexual risk
* Awareness of sexual and reproductive health services

ELIGIBILITY:
Inclusion Criteria:

* 9th grade student at a participating high school in East or South Los Angeles
* Written parent/guardian consent and student assent to participate

Exclusion Criteria:

* None

Ages: 13 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1909 (Actual)
Dates: Start 2011-09; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norman A. Constantine, PhD, Principal Investigator — Public Health Institute; Louise A. Rohrbach, PhD, MPH, Principal Investigator — University of Southern California
Locations (1):
- Planned Parenthood Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Constantine NA, Jerman P, Berglas NF, Angulo-Olaiz F, Chou CP, Rohrbach LA. Short-term effects of a rights-based sexuality education curriculum for high-school students: a cluster-randomized trial. BMC Public Health. 2015 Mar 26;15:293. doi: 10.1186/s12889-015-1625-5. PMID 25886554

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In Year 1 (2011-12), eight schools participated. Following the first year, one matched pair of schools dropped out due to school administration changes and a new matched pair of schools with similar student characteristics was added for Year 2 (2012-13). Thus, ten schools participated in intervention delivery over the study period.
Pre-assignment Details: 1909 participants were enrolled.
Period: Overall Study
Arm/Group | SEI Classroom Curriculum | Control Classroom Curriculum
Started | 1025 | 884
SEI Curriculum Only | 461 | 0
SEI Curriculum + 3 SchoolWide Components | 544 | 0
Ctrl Curriculum Only | 0 | 456
Ctrl Curriculm +1 SchoolWide Component | 0 | 428
Completed | 769 | 678
Not Completed | 256 | 206
Not completed — Lost to Follow-up | 256 | 206

BASELINE CHARACTERISTICS:
Population: Intervention groups were similar on baseline characteristics.
Groups:
- Total: Total of all reporting groups
Arm/Group | SEI Classroom Curriculum | Control Classroom Curriculum | Total
Number analyzed (Participants) | 1025 | 884 | 1909
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1025 | 884 | 1909
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.15 (.60) | 14.16 (.55) | 14.15 (.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 518 | 448 | 966
  Male | 507 | 436 | 943
Region of Enrollment [Number; unit: participants]
  United States | 1025 | 884 | 2881

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With Pregnancy Risk
Description: Between-arm difference in percent of youth who report engaging in recent sexual intercourse but not using birth control and/or condoms
Time Frame: 1 year
Population: 412 participants completed the SEI Curriculum + 3 School Wide Components Arm/Group and 329 completed the Control Curriculum + 1 School Wide Component Arm/Group. Small fractional inconsistencies in reported and calculated outcome results are due to missing data and/or rounding of percentages.
Measure: Number; unit: percentage of participants
Groups:
- SEI Curriculum + 3 School Wide Components: Participants receive SEI curriculum and three school wide components (peer advocacy and education, parent education, clinical services linkages).
  3 School Wide Components: Participants receive all three school wide components. The peer education and advocacy component recruits, trains and supervises students through an after-school leadership program to serve as resources to peers, organize health events, and refer students to school-based clinic services. The parent education component provides sessions for parents of students, covering reproductive health, teen pregnancy, and parent-teen communication, together with a parent education booklet for widespread use. This clinical services linkages includes "clinic without walls" health services on campus, including pregnancy/STI testing, contraceptive consultation and prescriptions, condom distribution, counseling, and referrals. It includes training for teachers and staff to distribute condoms as needed.
- Control Curriculum + 1 School Wide Component: Participants receive control curriculum and one of the three school wide components (clinical services linkages).
  1 School Wide Component: Participants receive one of the three school wide components, the clinical services linkages. This component includes "clinic without walls" health services on campus for students, including pregnancy and STI testing, contraceptive consultation and prescriptions, condom distribution, counseling, and referrals. It also includes training for teachers and school staff to distribute condoms to students as needed.
Arm/Group | SEI Classroom Curriculum | Control Classroom Curriculum | SEI Curriculum + 3 School Wide Components | Control Curriculum + 1 School Wide Component
Number analyzed (Participants) | 769 | 678 | 412 | 329
percentage of participants | 11.8 | 11.1 | 10.2 | 10.8
Statistical Analysis 1: Comparison: SEI Classroom Curriculum vs Control Classroom Curriculum; Test type: Superiority; p = 0.6430, Regression, Logistic; Multilevel model to account for classroom/school clusters. Adjusted for student/classroom gender, student/classroom sexual experience, pretest score; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.75 to 1.60]
Statistical Analysis 2: Comparison: SEI Curriculum + 3 School Wide Components vs Control Curriculum + 1 School Wide Component; Test type: Superiority; p = 0.3718, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.75, 95% CI 2-sided [0.39 to 1.44]

2. Primary Outcome: Percent of Participants With Sexually Transmitted Infection (STI) Risk
Description: Between-arm difference in percent of youth who report engaging in recent vaginal, anal and/or oral sexual intercourse but not using condoms
Time Frame: 1 year
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Groups:
- SEI Curriculum + 3 School Wide Components: Participants receive SEI classroom curriculum and three school wide components (peer advocacy and education, parent education, clinical services linkages).
  3 School Wide Components: Participants receive all three school wide components. The peer education and advocacy component recruits, trains and supervises students through an after-school leadership program to serve as resources to peers, organize health events, and refer students to school-based clinic services. The parent education component provides sessions for parents of students, covering reproductive health, teen pregnancy, and parent-teen communication, together with a parent education booklet for widespread use. This clinical services linkages includes "clinic without walls" health services on campus, including pregnancy/STI testing, contraceptive consultation and prescriptions, condom distribution, counseling, and referrals. It includes training for teachers and staff to distribute condoms as needed.
- Control Curriculum + 1 School Wide Component: Participants receive control classroom curriculum and one of the three school wide components (clinical services linkages).
  1 School Wide Component: Participants receive one of the three school wide components, the clinical services linkages. This component includes "clinic without walls" health services on campus for students, including pregnancy and STI testing, contraceptive consultation and prescriptions, condom distribution, counseling, and referrals. It also includes training for teachers and school staff to distribute condoms to students as needed.
Arm/Group | SEI Classroom Curriculum | Control Classroom Curriculum | SEI Curriculum + 3 School Wide Components | Control Curriculum + 1 School Wide Component
Number analyzed (Participants) | 769 | 678 | 412 | 329
percentage of participants | 12.8 | 13.4 | 11.0 | 13.8
Statistical Analysis 1: Comparison: SEI Classroom Curriculum vs Control Classroom Curriculum; Test type: Superiority; p = 0.8083, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.67 to 1.37]
Statistical Analysis 2: Comparison: SEI Curriculum + 3 School Wide Components vs Control Curriculum + 1 School Wide Component; Test type: Superiority; p = 0.1083, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.60, 95% CI 2-sided [0.32 to 1.13]

3. Primary Outcome: Percent of Participants With Multiple Sexual Partners
Description: Between-arm difference in percent of youth who report having more than one recent vaginal, anal and/or oral sexual partner
Time Frame: 1 year
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Groups:
- SEI Curriculum + 3 School Wide Components: Participants receive the SEI classroom curriculum and three school wide components (peer advocacy and education, parent education, clinical services linkages).
  3 School Wide Components: Participants receive all three school wide components. The peer education and advocacy component recruits, trains and supervises students through an after-school leadership program to serve as resources to peers, organize health events, and refer students to school-based clinic services. The parent education component provides sessions for parents of students, covering reproductive health, teen pregnancy, and parent-teen communication, together with a parent education booklet for widespread use. This clinical services linkages includes "clinic without walls" health services on campus, including pregnancy/STI testing, contraceptive consultation and prescriptions, condom distribution, counseling, and referrals. It includes training for teachers and staff to distribute condoms as needed.
- Control Curriculum + 1 School Wide Component: Participants receive the control curriculum and one school wide component (clinical services linkages).
  1 School Wide Component: Participants receive one of the three school wide components, the clinical services linkages. This component includes "clinic without walls" health services on campus for students, including pregnancy and STI testing, contraceptive consultation and prescriptions, condom distribution, counseling, and referrals. It also includes training for teachers and school staff to distribute condoms to students as needed.
Arm/Group | SEI Classroom Curriculum | Control Classroom Curriculum | SEI Curriculum + 3 School Wide Components | Control Curriculum + 1 School Wide Component
Number analyzed (Participants) | 769 | 678 | 412 | 329
percentage of participants | 4.3 | 5.6 | 2.9 | 5.8
Statistical Analysis 1: Comparison: SEI Classroom Curriculum vs Control Classroom Curriculum; Test type: Superiority; p = 0.1006, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.62, 95% CI 2-sided [0.35 to 1.10]
Statistical Analysis 2: Comparison: SEI Curriculum + 3 School Wide Components vs Control Curriculum + 1 School Wide Component; Test type: Superiority; p = 0.2117, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.49, 95% CI 2-sided [0.16 to 1.53]

4. Primary Outcome: Percent of Participants Who Ever Used Sexual and Reproductive Health Services
Description: Between-arm difference in percent of youth who report ever using sexual and reproductive health services
Time Frame: 1 year
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | SEI Classroom Curriculum | Control Classroom Curriculum | SEI Curriculum + 3 School Wide Components | Control Curriculum + 1 School Wide Component
Number analyzed (Participants) | 769 | 678 | 412 | 329
percentage of participants | 27.7 | 21.7 | 28.9 | 16.0
Statistical Analysis 1: Comparison: SEI Classroom Curriculum vs Control Classroom Curriculum; Test type: Superiority; p = 0.0218, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.37, 95% CI 2-sided [1.05 to 1.78]
Statistical Analysis 2: Comparison: SEI Curriculum + 3 School Wide Components vs Control Curriculum + 1 School Wide Component; Test type: Superiority; p = 0.0211, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.73, 95% CI 2-sided [1.09 to 2.75]

5. Secondary Outcome: Percent of Participants Who Ever Had Sex
Description: Between-arm difference in percent of youth who report ever engaging in vaginal and/or anal sexual intercourse
Time Frame: 1 year
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | SEI Classroom Curriculum | Control Classroom Curriculum | SEI Curriculum + 3 School Wide Components | Control Curriculum + 1 School Wide Component
Number analyzed (Participants) | 769 | 678 | 412 | 329
percentage of participants | 31.2 | 28.6 | 30.2 | 26.7
Statistical Analysis 1: Comparison: SEI Classroom Curriculum vs Control Classroom Curriculum; Test type: Superiority; p = 0.1763, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.90 to 1.73]
Statistical Analysis 2: Comparison: SEI Curriculum + 3 School Wide Components vs Control Curriculum + 1 School Wide Component; Test type: Superiority; p = 0.5869, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.85, 95% CI 2-sided [0.45 to 1.58]

6. Secondary Outcome: Percent of Participants Who Ever Had Oral Sex
Description: Between-arm difference in percent of youth who report ever engaging in oral sexual intercourse
Time Frame: 1 year
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | SEI Classroom Curriculum | Control Classroom Curriculum | SEI Curriculum + 3 School Wide Components | Control Curriculum + 1 School Wide Component
Number analyzed (Participants) | 769 | 678 | 412 | 329
percentage of participants | 22.2 | 22.6 | 21.3 | 23.9
Statistical Analysis 1: Comparison: SEI Classroom Curriculum vs Control Classroom Curriculum; Test type: Superiority; p = 0.8102, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.75 to 1.44]
Statistical Analysis 2: Comparison: SEI Curriculum + 3 School Wide Components vs Control Curriculum + 1 School Wide Component; Test type: Superiority; p = 0.2956, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.72, 95% CI 2-sided [0.39 to 1.34]

7. Secondary Outcome: Percent of Participants With Recent Sexual Activity
Description: Between-arm difference in percent of youth who report engaging in vaginal and/or anal sexual intercourse during the last 3 months
Time Frame: 1 year
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | SEI Classroom Curriculum | Control Classroom Curriculum | SEI Curriculum + 3 School Wide Components | Control Curriculum + 1 School Wide Component
Number analyzed (Participants) | 769 | 678 | 412 | 3
percentage of participants | 18.2 | 16.7 | 16.0 | 16.4
Statistical Analysis 1: Comparison: SEI Classroom Curriculum vs Control Classroom Curriculum; Test type: Superiority; p = 0.4645, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.13, 95% CI 2-sided [0.82 to 1.56]
Statistical Analysis 2: Comparison: SEI Curriculum + 3 School Wide Components vs Control Curriculum + 1 School Wide Component; Test type: Superiority; p = 0.3809, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.77, 95% CI 2-sided [0.43 to 1.40]

8. Secondary Outcome: Percent of Participants With Recent Oral Sex Activity
Description: Between-arm difference in percent of youth who report engaging in oral sexual intercourse in the last 3 months
Time Frame: 1 year
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | SEI Classroom Curriculum | Control Classroom Curriculum | SEI Curriculum + 3 School Wide Components | Control Curriculum + 1 School Wide Component
Number analyzed (Participants) | 769 | 678 | 412 | 329
percentage of participants | 10.7 | 13.0 | 9.3 | 14.2
Statistical Analysis 1: Comparison: SEI Classroom Curriculum vs Control Classroom Curriculum; Test type: Superiority; p = 0.1335, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.75, 95% CI 2-sided [0.52 to 1.09]
Statistical Analysis 2: Comparison: SEI Curriculum + 3 School Wide Components vs Control Curriculum + 1 School Wide Component; Test type: Superiority; p = 0.0741, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.56, 95% CI 2-sided [0.29 to 1.06]

9. Secondary Outcome: Percent of Participants Who Used Condom at Last Sex
Description: Between-arm difference in percent of youth who report using a condom the last time they had sexual intercourse
Time Frame: 1 year
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | SEI Classroom Curriculum | Control Classroom Curriculum | SEI Curriculum + 3 School Wide Components | Control Curriculum + 1 School Wide Component
Number analyzed (Participants) | 769 | 678 | 412 | 329
percentage of participants | 59.8 | 58.9 | 60.9 | 57.9
Statistical Analysis 1: Comparison: SEI Classroom Curriculum vs Control Classroom Curriculum; Test type: Superiority; p = 0.9085, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.54 to 2.01]
Statistical Analysis 2: Comparison: SEI Curriculum + 3 School Wide Components vs Control Curriculum + 1 School Wide Component; Test type: Superiority; p = 0.8059, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.36 to 3.62]

10. Secondary Outcome: Percent of Participants Who Used Contraceptive at Last Sex
Description: Between-arm difference in percent of youth who report using birth control and/or condoms the last time they had sexual intercourse
Time Frame: 1 year
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | SEI Classroom Curriculum | Control Classroom Curriculum | SEI Curriculum + 3 School Wide Components | Control Curriculum + 1 School Wide Component
Number analyzed (Participants) | 769 | 678 | 412 | 329
percentage of participants | 64.2 | 68.1 | 65.6 | 64.9
Statistical Analysis 1: Comparison: SEI Classroom Curriculum vs Control Classroom Curriculum; Test type: Superiority; p = 0.6861, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.87, 95% CI 2-sided [0.44 to 1.71]
Statistical Analysis 2: Comparison: SEI Curriculum + 3 School Wide Components vs Control Curriculum + 1 School Wide Component; Test type: Superiority; p = 0.9973, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 0 — No results provided, as model would not converge

11. Secondary Outcome: Percent of Participants Who Currently Have Condom
Description: Between-arm difference in percent of youth who report currently having a condom with them (e.g., in a pocket, purse or backpack)
Time Frame: 1 year
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | SEI Classroom Curriculum | Control Classroom Curriculum | SEI Curriculum + 3 School Wide Components | Control Curriculum + 1 School Wide Component
Number analyzed (Participants) | 769 | 678 | 412 | 329
percentage of participants | 18.4 | 10.4 | 20.3 | 9.3
Statistical Analysis 1: Comparison: SEI Classroom Curriculum vs Control Classroom Curriculum; Test type: Superiority; p = 0.0002, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.97, 95% CI 2-sided [1.39 to 2.80]
Statistical Analysis 2: Comparison: SEI Curriculum + 3 School Wide Components vs Control Curriculum + 1 School Wide Component; Test type: Superiority; p = 0.0030, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 2.71, 95% CI 2-sided [1.44 to 5.09]

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | SEI Classroom Curriculum | Control Classroom Curriculum | SEI Curriculum + 3 School Wide Components | Control Curriculum + 1 School Wide Component
All-Cause Mortality (participants affected / at risk) | 0/1025 | 0/884 | 0/544 | 0/428
Serious Adverse Events (participants affected / at risk) | 0/1025 | 0/884 | 0/544 | 0/428
Other Adverse Events (participants affected / at risk) | 0/1025 | 0/884 | 0/544 | 0/428

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No